CLINICAL TRIAL: NCT05767749
Title: Characterizing and Comparing the Duration of Local Anesthetic in Dermatologic Surgery
Brief Title: Split Face Study of the Duration of Local Anesthetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-10025244
Record Dates: First submitted 2023-02-22; First posted 2023-03-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Anesthetics, Local
Keywords: Anesthesia; Mohs; lidocaine; ropivacaine; bupivacaine
MeSH Terms: interventions — Lidocaine; Epinephrine; Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 0.5mL of local anesthetic will be injected into the skin of each participant by the one dermatologic surgeon (PI of the study, Dr. Kira Minkis, KM). Dr. Minkis will be unblinded to the laterality of the anesthetics and will not be involved in further assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lidocaine + epinephrine vs Ropivacaine (Experimental): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed. Participants in this arm will receive an injection of 0.5ml of . Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into one side of the nose (nasal ala) and 0.5ml of Naropin (ropivacaine) 0.5% into the opposite nasal ala. Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes on both sides of the face, until the patient reports return of a sharp sensation upon the pinprick test.
  Interventions: Drug: lidocaine + epinephrine 1:100,000; Drug: Ropivacaine 0.5% Injectable Solution
- Lidocaine + epinephrine vs Bupivacaine (Experimental): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed. Participants in this arm will receive an injection of 0.5ml of lidocaine + epinephrine into one side of the nose (nasal ala) and 0.5ml of Marcaine (bupivacaine) 0.5% into the opposite nasal ala. Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes on both sides of the face, until the patient reports return of a sharp sensation upon the pinprick test.
  Interventions: Drug: lidocaine + epinephrine 1:100,000; Drug: Bupivacaine 0.5% Injectable Solution
- Ropivacaine vs Bupivacaine (Experimental): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed. Participants in this arm will receive an injection of 0.5ml of Naropin (ropivacaine) 0.5% into one side of the nose (nasal ala) and 0.5ml of Marcaine (bupivacaine) 0.5% into the opposite nasal ala. Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes on both sides of the face, until the patient reports return of a sharp sensation upon the pinprick test.
  Interventions: Drug: Ropivacaine 0.5% Injectable Solution; Drug: Bupivacaine 0.5% Injectable Solution

INTERVENTIONS:
Drug: lidocaine + epinephrine 1:100,000 — 0.5 ml lidocaine + epinephrine 1:100,000, buffered 1/10 with sodium bicarb.
  Other Names: Xylocaine + epinephrine 1:100,000
  Arms: Lidocaine + epinephrine vs Bupivacaine; Lidocaine + epinephrine vs Ropivacaine
Drug: Ropivacaine 0.5% Injectable Solution — 0.5 ml Ropivacaine 0.5% Injectable Solution
  Other Names: Naropin
  Arms: Lidocaine + epinephrine vs Ropivacaine; Ropivacaine vs Bupivacaine
Drug: Bupivacaine 0.5% Injectable Solution — 0.5ml bupivacaine 0.5%
  Other Names: Marcaine
  Arms: Lidocaine + epinephrine vs Bupivacaine; Ropivacaine vs Bupivacaine

SUMMARY:
This is a research study to compare how long injectable pain medications (anesthetics) commonly used in dermatologic surgery are effective for. This study will compare a short-acting anesthetic, lidocaine with epinephrine, to one of two long-acting anesthetics (ropivacaine or bupivacaine). This study will also directly compare the duration of actions of ropivacaine and bupivacaine. The investigators hypothesize that the duration of anesthesia of short-acting anesthetics will not differ significantly from long-acting anesthetics at a single site and there will not be a significant difference between the two long-acting anesthetics at a single site.

DETAILED DESCRIPTION:
This study will compare the relative durations of local anesthetics within the same subject at a highly vascularized anatomic region of skin, the nasal ala. This study will test and compare the relative durations and efficacy of commonly used long acting (ropivacaine or bupivacaine) and short acting local anesthetics (lidocaine with epinephrine), delivered via local anesthesia. This study will use a modification of a previously published approach of non-invasive pinprick testing to assess the duration of local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Normal skin sensation at both nasal ala assessed by pinprick
* Ability to provide informed consent

Exclusion Criteria:

* Previous adverse reaction to local anesthetic or any components of the local anesthetics being evaluated
* Pregnant or breastfeeding volunteers (assessed by self-report)
* Patients taking monoamineoxidase inhibitors (MAOI) or antidepressants of the triptyline or imipramine types

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kira Minkis, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 subjects were recruited from March to July, 2023 at one site.
Units Other Than Participants: nasal ala
Groups:
- Lidocaine+Epinephrine (vs Ropivacaine): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed.
  Participants in this arm will receive an injection of 0.5ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into one side of the nose (nasal ala) (compared to 0.5ml of Naropin (ropivacaine) 0.5% into the opposite nasal ala).
  Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes , until the patient reports return of a sharp sensation upon the pinprick test.
  Agent: lidocaine + epinephrine 1:100,000: 0.5 ml lidocaine + epinephrine 1:100,000, buffered 1/10 with sodium bicarb.
- Ropivacaine (vs Lidocaine+Epinephrine): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed.
  Participants in this arm will receive an injection of 0.5ml of Naropin (ropivacaine) 0.5% into one side of the nose (nasal ala) (compared to 0.5ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into the opposite nasal ala).
  Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes , until the patient reports return of a sharp sensation upon the pinprick test.
  Agent: Ropivacaine 0.5% Injectable Solution: 0.5 ml Ropivacaine 0.5% Injectable Solution
- Lidocaine+Epinephrine (vs Bupivacaine): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed.
  Participants in this arm will receive an injection of 0.5ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into one side of the nose (nasal ala) (compared to 0.5ml bupivacaine 0.5% into the opposite nasal ala).
  Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes , until the patient reports return of a sharp sensation upon the pinprick test.
  Agent: lidocaine + epinephrine 1:100,000: 0.5 ml lidocaine + epinephrine 1:100,000, buffered 1/10 with sodium bicarb.
- Bupivacaine (vs Lidocaine+Epinephrine): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed.
  Participants in this arm will receive an injection of 0.5ml bupivacaine 0.5% into one side of the nose (nasal ala) (compared to 0.5ml of Xylocaine + epinephrine 1:100,000 (lidocaine + epinephrine 1:100,000), buffered 1/10 with sodium bicarb into the opposite nasal ala).
  Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes , until the patient reports return of a sharp sensation upon the pinprick test.
  Agent: Bupivacaine 0.5% Injectable Solution: 0.5ml bupivacaine 0.5%
- Ropivacaine (vs Bupivacaine): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed.
  Participants in this arm will receive an injection of 0.5 ml Ropivacaine 0.5% into one side of the nose (nasal ala) (compared to 0.5ml bupivacaine 0.5% into the opposite nasal ala).
  Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes , until the patient reports return of a sharp sensation upon the pinprick test.
  Agent: Ropivacaine 0.5% Injectable Solution: 0.5 ml Ropivacaine 0.5% Injectable Solution
- Bupivacaine (vs Ropivacaine): Each site of the nasal ala will be tested for normal sensation using sterile 30-gauge needles. Other eligibility criteria will be confirmed.
  Participants in this arm will receive an injection of 0.5ml bupivacaine 0.5% into one side of the nose (nasal ala) (compared to 0.5 ml Ropivacaine 0.5% into the opposite nasal ala).
  Laterality of each anesthetic administration will be randomly assigned for each patient. Subjects will be evaluated for duration of effect of anesthesia every 15 minutes , until the patient reports return of a sharp sensation upon the pinprick test.
  Agent: Bupivacaine 0.5% Injectable Solution: 0.5ml bupivacaine 0.5%
Period: Overall Study
Arm/Group | Lidocaine+Epinephrine (vs Ropivacaine) | Ropivacaine (vs Lidocaine+Epinephrine) | Lidocaine+Epinephrine (vs Bupivacaine) | Bupivacaine (vs Lidocaine+Epinephrine) | Ropivacaine (vs Bupivacaine) | Bupivacaine (vs Ropivacaine)
Started | 24; 24 nasal ala | 24; 24 nasal ala | 25; 25 nasal ala | 25; 25 nasal ala | 26; 26 nasal ala | 26; 26 nasal ala
Completed | 24; 24 nasal ala | 24; 24 nasal ala | 23; 23 nasal ala | 23; 23 nasal ala | 24; 24 nasal ala | 24; 24 nasal ala
Not Completed | 0; 0 nasal ala | 0; 0 nasal ala | 2; 2 nasal ala | 2; 2 nasal ala | 2; 2 nasal ala | 2; 2 nasal ala
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants were excluded from analysis if they withdrew from the study (1 participant), did not regain sensation bilaterally before leaving the study site (3 participants), or, if the time to regain sensation could not be accurately determined (1 participant).
Units Other Than Participants: nasal ala
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine+Epinephrine (vs Ropivacaine) | Ropivacaine (vs Lidocaine+Epinephrine) | Lidocaine+Epinephrine (vs Bupivacaine) | Bupivacaine (vs Lidocaine+Epinephrine) | Ropivacaine (vs Bupivacaine) | Bupivacaine (vs Ropivacaine) | Total
Number analyzed (Participants) | 24 | 24 | 25 | 25 | 26 | 26 | 75
Number analyzed (nasal ala) | 23 | 23 | 23 | 23 | 24 | 24 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 6 | 6 | 6 | 6 | 44
  >=65 years | 14 | 14 | 19 | 19 | 20 | 20 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 8 | 8 | 10 | 10 | 54
  Male | 15 | 15 | 17 | 17 | 16 | 16 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 0 | 0 | 4
  Not Hispanic or Latino | 24 | 24 | 23 | 23 | 24 | 24 | 142
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 22 | 22 | 22 | 22 | 23 | 23 | 134
  More than one race | 1 | 1 | 0 | 0 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 2 | 2 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Return to Baseline Sensation, as Determined by Binary Outcomes (Yes/no) in 15 Minute Increments
Description: To determine whether the time to return to baseline sensation differs significantly between each pair of anesthetics, the investigators will measure the time to return to baseline sensation at each anesthetized site by asking participants at 15 minute intervals if they can feel a sharp sensation at the site. Sterile needles will be used. The return of the sensitivity will be determined using binary outcomes (yes/no) and recorded on a standardized template. The maximum difference in anesthetic duration that the investigators consider "not different" from a clinical standpoint is 15 minutes.
Time Frame: Up to 4 hours.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Minutes
Units Other Than Participants: nasal Ala
Arm/Group | Lidocaine+Epinephrine (vs Ropivacaine) | Ropivacaine (vs Lidocaine+Epinephrine) | Lidocaine+Epinephrine (vs Bupivacaine) | Bupivacaine (vs Lidocaine+Epinephrine) | Ropivacaine (vs Bupivacaine) | Bupivacaine (vs Ropivacaine)
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 24 | 24
Number analyzed (nasal Ala) | 23 | 23 | 23 | 23 | 24 | 24
Minutes | 54.34 (27.48) | 49.86 (22.53) | 43.13 (22.20) | 55.78 (24.62) | 52.33 (24.09) | 46.16 (20.24)
Statistical Analysis 1: Comparison: Lidocaine+Epinephrine (vs Ropivacaine) vs Lidocaine+Epinephrine (vs Bupivacaine); Test type: Superiority; p = 0.93, t-test, 2 sided; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-12.8 to 14.0] — Direction = (Lidocaine + epinephrine vs Ropivacaine) minus (Lidocaine + epinephrine vs Bupivacaine)
Statistical Analysis 2: Comparison: Lidocaine+Epinephrine (vs Ropivacaine) vs Ropivacaine (vs Bupivacaine); Test type: Superiority; p = 0.54, t-test, 2 sided; Mean Difference (Final Values) = 3.73, 95% CI 2-sided [-8.3 to 15.8] — Direction = (Lidocaine + epinephrine vs Ropivacaine) minus (Ropivacaine vs Bupivacaine)
Statistical Analysis 3: Comparison: Lidocaine+Epinephrine (vs Bupivacaine) vs Ropivacaine (vs Bupivacaine); Test type: Superiority; p = 0.60, t-test, 2 sided; Mean Difference (Final Values) = 3.12, 95% CI 2-sided [-8.7 to 15.0] — Direction = (Lidocaine + epinephrine vs Bupivacaine) minus (Ropivacaine vs Bupivacaine)

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events for the duration of their study visit (1 day).
Arm/Group | Lidocaine+Epinephrine (vs Ropivacaine) | Ropivacaine (vs Lidocaine+Epinephrine) | Lidocaine+Epinephrine (vs Bupivacaine) | Bupivacaine (vs Lidocaine+Epinephrine) | Ropivacaine (vs Bupivacaine) | Bupivacaine (vs Ropivacaine)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/25 | 0/25 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/25 | 0/25 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/25 | 0/25 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05767749/Prot_SAP_000.pdf